CLINICAL TRIAL: NCT02541136
Title: Neural and Stress Correlates of Resilience in an Exercise-behavioural Programme
Brief Title: Neural Changes of Exercise: a Functional MRI Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Thomas Frodl, Professor, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Rec Ref 2011/45/13
Record Dates: First submitted 2015-08-28; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Aerobic Exercise
Keywords: exercise; resilience; physiotherapy; fMRI
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental): Participants in this arm took part in the aerobic exercise component of the study and attended St. James's Hospital in Dublin twice a week for 16 weeks. Furthermore, exercising participants were asked to engage in recorded aerobic activity outside of the class, which followed a standardised progression from 1-3 additional sessions, at the same intensity as the week's class.
  Interventions: Behavioral: Aerobic Exercise
- Control (No Intervention): Participants in the control group didn't change their sedentary habits.

INTERVENTIONS:
Behavioral: Aerobic Exercise — Each exercise class consisted of a warm-up, an aerobic and a cool-down phase, supervised by a physiotherapist. The warm up and cool down phases consisted of 5-7 minutes of low intensity aerobic exercise, < 40% Heart Rate Reserve (HHR), to allow the cardiopulmonary and musculoskeletal systems to adapt and recover, respectively.
  The aerobic component initially consisted of 21 minutes at an intensity of 40-59% HRR and was progressed to 42 minutes at 55-75% HRR by week 8 until programme completion. All participants worked at the same intensity and duration at the various time points throughout the study. Continuous, rhythmic exercise using large muscle groups was prescribed using treadmills, cycle ergometers and other aerobic exercise that increased heart rate to its prescribed level.
  Arms: Exercise

SUMMARY:
Stress-related disorders have a profound impact on public health. The World Health Organisation (WHO) found major depressive disorder (MDD) to be one of the most important human health problems with a prevalence of about 10%. In the current proposal the aim is to investigate mechanisms of resilience against stress-related disorders and to examine changes in quality of life, health, brain structure and brain function in individuals performing a "resilience" programme. Therefore, the investigators will recruit forty healthy subjects from the hospital staff exposed to "normal" day-to-day stress and not participating already in a fitness programme. Half of the subjects will be randomised to a cognitive behavioural self-experience and exercise programme for 20 weeks carried out by experienced supervisors, coaches and trainers. Clinical psychological and psychiatric examinations will be carried out weekly and a range of sophisticated neuroimaging techniques - high angular resolution diffusion imaging (HARDI) and functional MRI (fMRI) - will be conducted before and after the "resilience" program in order to investigate its effectiveness on brain structure and function. The stress system will also be tested by examining cortisol awaking response (CAR) and daily rhythms of cortisol secretion. These techniques are all well established in our laboratories. The proposed research will likely stimulate the development of new prevention strategies for this common and important disorder, and in the future could be applied to other illnesses. Moreover, when successful it could be patented and offered for implementation in the daily routine of median to large companies.

DETAILED DESCRIPTION:
Mental disorders are a major cause of long-term disability and are a direct cause of mortality, with approximately 800,000 individuals dying from suicide every year worldwide - a high proportion of them arise from major depressive disorder (MDD). Knowledge of MDD has expanded in recent years by detecting that neuroplasticity may play a core role in the pathophysiology of the disease. Neuroplasticity in this context refers to the brain's ability to change and thus might be the presupposition for building up strategies against mental disorders.

The best-characterized and most studied examples of neuroplasticity are the molecular and cellular adaptations underlying learning and exercise. Exercise improves cognition, has antidepressant effects and was also found to have positive effects on the brain structure as measured with magnetic resonance imaging (MRI). Further, research in older adults indicates that increased aerobic fitness can be neuroprotective and can enhance brain structure and function. Increase of gray matter volume in parietal and frontal brain regions and corresponding increases of diffusivity in white matter fibres were seen as early as after 2 weeks of training a balancing task.

On the other hand experimental studies found that stress and chronic exposure to high levels of glucocorticoids leads to depressive-like states. These states were accompanied by atrophy and loss of neurons in the adult hippocampus which is a temporal lobe brain region involved in learning, memory and mood regulation. Hippocampal damage, resulting from excessive exposure of the brain to glucocorticoids, leads to impaired feedback inhibition of hypothalamic-pituitary-adrenal (HPA) axis by glucocorticoids, causing unrestrained release of the axis - the "Glucocorticoid Cascade Hypothesis". Prolonged stress, or an excess allostatic load, is thus harmful and is probably important in the processes mediating dementias. Efficient stress responses are necessary to cope with changes in the environment and an ability to terminate the stress response is of central importance in the return to homeostasis. Individuals with depression have relatively high cortisol secretory tone with blunted diurnal secretory patterns of cortisol secretion, reflecting poor regulatory feedback in the hippocampus. Higher cortisol stress responses to awakening (CAR), conversely, are found in those who are chronically stressed, depressed or remitted from depression or bipolar disorder, and in adolescents who will later develop depression.

Interestingly, the investigators found that structural changes of the hippocampus, a brain region involved in memory and emotion regulation, become more pronounced when a patient with depression develops a chronic disease course. Recently, they detected that hippocampal volumes from patients with MDD, who carry also a genetic risk-allele (SLC6A4, 5-HTTLPR), were smaller when they had a history of emotional neglect compared to patients who had only the genetic or the emotional neglect risk factor separately. In the context of neuroimaging, diffusion tensor imaging (DTI), which is a significant step forward for characterizing microstructural changes or differences, is highly interesting. Using high angular resolution diffusion imaging, the investigators found that unaffected healthy first degree relatives of patients with MDD with stronger fiber connections between prefrontal and temporo-parietal brain regions managed incidences of early life adversity without later developing depression suggesting that resilience may be associated with stronger connections. This line of research suggests that structural and functional brain changes are already there before the manifestation of the disease and that these changes seem to be related to the individuals' vulnerability.

Thus, preventing these brain changes, normalizing the stress functions and increasing the resilience of individuals is a major challenge for the future in order to prevent major stress-related mental disorders. The ability of the brain to adapt suggests that it might be possible to increase resilience in order to protect an individual from becoming depressed. In addition to exercise and learning, cognitive behavioral therapy (CBT) and remediation programs have been shown to have effects on brain structure and function in patients with manifest disorders like depression or schizophrenia and especially the combination of CBT with exercise and learning might result in most prominent outcomes. Neuroplastic brain changes have been reported with CBT. For example, behavioral activation therapy for depression, a psychotherapy modality designed to increase engagement with positive stimuli and reduce avoidance behaviors, resulted in decreased activations in prefrontal structures, including the paracingulate gyrus, the right orbitofrontal cortex, and the right frontal pole, while symptoms of depression improved. Elevated amygdala-hippocampal activity decreased and reduced ACC activity increased during 16 weeks of CBT in 16 patients with MDD. A recent review highlights the effects of brief working memory training across different studies on brain activation in multiple regions including the dorsolateral prefrontal cortex, parietal cortex, and occipital cortex. Interestingly, cycling has been shown to increase the volume of the hippocampus in both patients with schizophrenia and healthy comparison subjects, with no change in the non-exercise group of patients. This suggests that CBT and exercise can have an impact on the recovery of the brain system from conditions like schizophrenia and MDD.

Effects of a resilience program have never been investigated with neuroimaging, although it would be possible to achieve information about the structure of the white matter fiber bundles that connect certain brain regions. Psychological constructs that promote resilience - the ability to cope with stressful situations - include commitment, patience, optimism and self-esteem, in addition to the capacity to modulate emotions and to develop adaptive social behavior. These traits implicate the brain's cognitive-emotional interplay, which seems to be a critical determinant of the emergence of pathological rather than resilient phenotypes. The cognitive-emotional interplay and its functional brain connectivity can be studied using functional MRI. Interestingly, using functional MRI it has been shown that a bias between emotional and cognitive processing exists in patients with MDD.

Aims:

The aim of the current proposal is to carry out a 20 weeks lasting extensive resilience program in order to stimulate resilience in a healthy unaffected population that is exposed to normal day-to-day work stress in the hospital. The investigators will measure the effectiveness of this program by examining behavioral, diurnal cortisol secretion rhythms and stress responses, microstructural as well as functional neural changes.

Hypotheses:

The "Resilience" program stimulates resilience indicated by

1. improved mood stability, better sleep quality and higher life quality
2. increase of hippocampal and anterior cingulate cortex volumes
3. increase of functional connectivity between frontal and limbic brain regions.
4. increase of fractional anisotropy (FA), which is a measure for the functioning of white matter fibers, between limbic and frontal brain regions.
5. increased gradient of the diurnal secretion in cortisol; and decrease in stress responses as measured by the cortisol awakening response

Methods and Materials Participants Forty healthy volunteers, e.g. from Adelaide and Meath Hospital, Dublin (AMiNCH) staff, will be recruited. They will have no history of neurological, mental (axis I and axis II) or chronic internal diseases. Further exclusion criteria for all participants will be a previous head injury with loss of consciousness. Moreover, they will not be members of fitness clubs or engage in intensive day to day activity. The 40 healthy volunteers will be randomized to a 20 week "resilience" program, 45 minutes exercise two times per week under the supervision of a physiotherapist as well as 2 home session; or to a control group without this program, and a further two sessions of 45-minute exercise/jogging will be completed each week Clinical assessments will be done weekly. Neuroimaging and salivary cortisol awaking tests will be carried out at baseline and after 20 weeks for both the resilience program group (N=20) and the control group (N=20).

Clinical assessments The NEO-FFI personality questionnaire and structured clinical interview for DSM disorders (SCID)-I and II will be carried out initially to exclude and history of, or current, psychiatric disorder. Mood will be assessed using the Hamilton Depression Rating Scale (HDRS), the Hamilton Anxiety Rating Scale (HAM-A), and the Beck Depression Inventory (BDI) at baseline and then bi-weekly. Moreover, current life stressors will be evaluated in an interview conducted according to Keller et al. on a weekly basis; Life quality (Study-Short Form 36-Item Health Survey (SF-36, QoL-Bref) and the Pittsburgh sleep quality index (PSQI), will also be carried out bi-weekly. Early life stress will be assessed using the childhood trauma questionnaire (CTQ). The NEO-FFI personality questionnaire and SCID-I and II will also be carried out at inclusion once. Handedness will be determined by the Edinburgh inventory.

Neuroimaging techniques MRI images will be obtained with a 3.0 Tesla MRI (Phillips Achieva), located in the Trinity College Institute of Neuroscience (TCIN). MRI will be carried out using a 60 minutes imaging protocol.

Diffusion Tensor Imaging (DTI): In vivo DTI will be acquired using a single-shot echo-planar imaging (EPI) sequence with SENSE parallel imaging scheme (SENSivitiy Encoding). The diffusion weighting will be encoded in 61 independent directions. After pre-processing in the program ExploreDTI, tractography with ExploreDTI and tract-based spatial statistics using TBSS (www.fmrib.ox.ac.uk/fsl/tbss/index.html, FSL) will be carried out. We have experience in using these technique and performing the analyses (25).

Functional MRI: In order to identify functional changes in the emotion regulation system, we will apply an fMRI paradigm. We will use an Echo Planar Imaging (EPI), T2*-weighted gradient-echo imaging to visualise BOLD contrast (TR 2000 ms, TE 30 ms, flip angle of 90°, matrix 80 x 80, FOV 224 x 224 x 150 mm, resolution: 3.5 x 3.5 mm, slice thickness: 3.5 mm). A cognitive-emotional inhibition task, which is well established in our laboratory, will be used. Participants will be asked to process visual emotional stimuli either in emotional or cognitive way. This task is chosen specifically, because it is known to elicit activity in prefrontal cortex, amygdala, gyrus cinguli, orbitofrontal cortex, regions implicated in the pathophysiology of MDD. SPM8-based standard analysis, functional connectivity analysis (33) and Psycho-Physiological Interaction (PPI) analysis will be done.

Structural techniques: Additionally, the aim is to track any structural changes and to confirm as well as extend recent findings in this area. Therefore, all subjects will be scanned with a T1-weighted 3D-MPRAGE sequence (repetition time, 8.5 ms; echo time, 3.5 ms; total acquisition time, 7 min 30 sec; number of acquisitions, 1; field of view, 250 x 256 x 160 mm; resolution: 0.86x0.86x0.86 mm). Region of interest (ROI) analysis of the hippocampus and amygdala as well as optimised voxel-based morphometry (VBM) will be used for data analysis as previously done in our lab.

Saliva cortisol samples These will be collected by participating subjects on two successive week-days, or working days. Subjects spit into a small plastic tube at wakening, and 30, 45, 60 and 90 min later; and in the evening (12h after waking) and just prior to going to bed. The samples can be stored by participants in a domestic fridge and posted in batch in a prepared envelope to the research centre.

Calculation of sample size The investigators have previously conducted a number of longitudinal imaging studies. Based on these experiences, 20 subjects in each group should be more than sufficient to obtain significant effects, where signal changes in the order of 0.2% to 0.3% are typically found in cognitive-emotional tasks or at least 5 % microstructural changes should be found in structural MRI or DTI. Thus, with 20 subjects the effects should be detectable.

ELIGIBILITY:
Inclusion Criteria

* healthy participants

Exclusion Criteria:

* MRI exclusion criteria like metal implants, pacemakers
* internal or neurological disorders
* substance or alcohol abuse
* substance or alcohol dependency in the past
* cortisol therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-10; Primary Completion 2014-10 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Resting state functional MRI | 16 weeks
  Magnetic resonance images from each participant were obtained with a Philips Achieva MRI scanner (Philips Medical System, Veenphuis 4-6, 5684 PC Best, The Netherlands) operating at 3 Tesla. The functional images were collected in single runs using a gradient echo (TE=28ms; TR=2000; field of view=131mm, flip angle=90°) sensitive to blood oxygenation level-dependent (BOLD) contrast (T2* weighting). A total of 37 contiguous 3.2 mm-thick slices were acquired parallel to the anterior posterior commissure plane (3mm approximately isotropic resolution), providing complete brain coverage. The fMRI run included 220 volumes acquired continuously lasting 7.2 min in total. Structural data (for definitive atlas transformation) included a high resolution sagittal, 3D T1-weighted Turbo Gradient Echo Sequence (TE=3.9ms, TR=8.5ms, TI=1060ms, flip angle=8°), 256×240 acquisition matrix, 1×1×1 mm voxels) scan.
  Resting state data were analysed using the software programs SPM8 and CONN

SECONDARY OUTCOMES:
Questionnaire for mental well being | 16 weeks
  Mental mood state (both are self-rating instruments) was assessed with the Profile of Mood States questionnaire. The Profile of Mood States (POMS) original scale contains 65 self-report items using the 5-point Likert Scale. Participants can choose from 0-4.
Questionnaire on physical activity | 16 weeks
  Physical activity outside of the programme, such as walking to work or similar, was assessed with the International Physical Activity Questionnaire (IPAQ). This questionnaire rates 5 different activities and time of activity is given in minutes/hours.
Questionnaire on physical health | 16 weeks
  Physical health was assessed with the SF 36-Item Health Survey. SF-36 is a set of generic, coherent, and easily administered quality-of-life self reported measures. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. To calculate the scores it is necessary to purchase special software. Pricing depends on the number of scores that the researcher needs to calculate.
  The eight sections are:
  vitality physical functioning bodily pain general health perceptions physical role functioning emotional role functioning social role functioning mental health

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Frodl, MD, Principal Investigator — University of Dublin, Trinity College

REFERENCES:
- [Background] Prince M, Patel V, Saxena S, Maj M, Maselko J, Phillips MR, Rahman A. No health without mental health. Lancet. 2007 Sep 8;370(9590):859-77. doi: 10.1016/S0140-6736(07)61238-0. PMID 17804063
- [Background] Duman RS. Pathophysiology of depression: the concept of synaptic plasticity. Eur Psychiatry. 2002 Jul;17 Suppl 3:306-10. doi: 10.1016/s0924-9338(02)00654-5. PMID 15177086
- [Background] Frodl TS, Koutsouleris N, Bottlender R, Born C, Jager M, Scupin I, Reiser M, Moller HJ, Meisenzahl EM. Depression-related variation in brain morphology over 3 years: effects of stress? Arch Gen Psychiatry. 2008 Oct;65(10):1156-65. doi: 10.1001/archpsyc.65.10.1156. PMID 18838632
- [Background] Frodl T, Reinhold E, Koutsouleris N, Donohoe G, Bondy B, Reiser M, Moller HJ, Meisenzahl EM. Childhood stress, serotonin transporter gene and brain structures in major depression. Neuropsychopharmacology. 2010 May;35(6):1383-90. doi: 10.1038/npp.2010.8. Epub 2010 Feb 10. PMID 20147891
- [Background] Dichter GS, Felder JN, Smoski MJ. The effects of Brief Behavioral Activation Therapy for Depression on cognitive control in affective contexts: An fMRI investigation. J Affect Disord. 2010 Oct;126(1-2):236-44. doi: 10.1016/j.jad.2010.03.022. Epub 2010 Apr 24. PMID 20421135
- [Background] Frodl T, Bokde AL, Scheuerecker J, Lisiecka D, Schoepf V, Hampel H, Moller HJ, Bruckmann H, Wiesmann M, Meisenzahl E. Functional connectivity bias of the orbitofrontal cortex in drug-free patients with major depression. Biol Psychiatry. 2010 Jan 15;67(2):161-7. doi: 10.1016/j.biopsych.2009.08.022. PMID 19811772
- [Derived] Frodl T, Strehl K, Carballedo A, Tozzi L, Doyle M, Amico F, Gormley J, Lavelle G, O'Keane V. Aerobic exercise increases hippocampal subfield volumes in younger adults and prevents volume decline in the elderly. Brain Imaging Behav. 2020 Oct;14(5):1577-1587. doi: 10.1007/s11682-019-00088-6. PMID 30927200